CLINICAL TRIAL: NCT00517738
Title: Impact and Safety of a Physical Training Program on Health-related Quality of Life in Patients With Cirrhosis and Portal Hypertension
Brief Title: Effect of Physical Training Program on Health-related Quality of Life in Cirrhosis
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran (Other)
Collaborators: Instituto Nacional de Cardiologia Ignacio Chavez (Other)
Responsible Party: Principal Investigator, Andres Duarte-Rojo, MD, PhD, Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran
Allocation: Randomized | Model: Parallel | Masking: None
Other Study IDs: CIIBH-Ref.1639/GAS 166-09/11-1
Record Dates: First submitted 2007-08-16; First posted 2007-08-17 (Estimated); Last update posted 2015-10-08 (Estimated); Status verified 2015-10

CONDITIONS: Cirrhosis
MeSH Terms: conditions — Fibrosis | interventions — Physical Conditioning, Human; Exercise; Nutrition Therapy; Diet

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Physical training - No encephalopathy (Experimental): Patients randomized to the physical training program and diet intervention
  Interventions: Other: Physical training; Other: Diet intervention
- Control - No encephalopathy (Active Comparator): Patients not allocated to exercise program, but undergoing diet intervention
  Interventions: Other: Diet intervention
- Physical training - Early encephalopathy (Experimental): Patients with early hepatic encephalopathy (minimal or clinical grade 1-2) randomized to the physical training program
  Interventions: Other: Physical training; Other: Diet intervention
- Control - Early encephalopathy (Active Comparator): Patients with early hepatic encephalopathy (minimal or clinical grades 1-2) not allocated to the physical training program, but undergoing diet intervention
  Interventions: Other: Diet intervention

INTERVENTIONS:
Other: Physical training — A program of exercising under strict surveillance, with endurance and coordination maneuvers
  Other Names: Exercise; Muscle ammonia metabolism
  Arms: Physical training - Early encephalopathy; Physical training - No encephalopathy
Other: Diet intervention — Energy intake tailored to basal metabolism and level of physical activity. Protein and sodium intake will be adjusted to 1.2-1.5 g/kg/d, and 1.5-2 g/d of salt, respectively. The latter will be adjusted only in those patients presenting ascites and/or edema
  Other Names: Nutritional therapy; Diet

SUMMARY:
Physical training improves quality of life (QOL) in non-hepatic diseases. It is possible that the same effect happens in patients with cirrhosis and portal hypertension. Hepatic encephalopathy may also benefit from physical activity by increasing ammonia metabolism. The intention of this study is to assess if patients can improve their QOL and hepatic encephalopathy during a physical training program, and to address its safety.

DETAILED DESCRIPTION:
Patients with cirrhosis and portal hypertension experience a marked deterioration in health-related quality of life (QOL), as it has been shown with the use of questionnaires such as Short-Form-36 (SF-36) and Chronic Liver Disease Questionnaire (CLDQ). The deterioration in QOL is progressively accentuated as liver failure advances. There is a positive association between the level of physical activity and the sense of QOL, and physical training programs have proved to be useful in improving QOL in cardiovascular and pulmonary diseases, and in conditions affecting cognition. Thereby, it is hypothesized that a physical training program may improve QOL and hepatic encephalopathy in patients with cirrhosis and portal hypertension. Data supporting physical activity as a way to improve hepatic encephalopathy derives from experimental models showing that skeletal muscle is able to remove blood ammonia, presumably by inducing the enzyme glutamine synthetase. However, it is uncertain whether such a program is safe, or if it can lead to an increase in portal hypertension and progression of the disease.

ELIGIBILITY:
Inclusion Criteria:

* Biopsy-proven or clinically evident cirrhosis
* Able to perform exercise

Exclusion Criteria:

* Overt hepatic encephalopathy grades 3 or 4
* Cardiovascular complications (pulmonary hypertension, heart failure)
* Diabetes mellitus and microangiopathic complications, or under treatment with insulin
* Renal failure
* Portal hypertension with high risk for variceal bleeding
* Hepatocellular carcinoma

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 29 (Actual)
Dates: Start 2007-02; Primary Completion 2014-01 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Improvement in QOL questionnaires | 3 months
  QOL will be measured by means of SF-36 and CLDQ
Lack of deterioration in portal hypertension | 3 months
  This will be measured by the hepatic vein pressure gradient (HVPG) through liver catheterization

SECONDARY OUTCOMES:
Improvement in cognitive status | 3 months
  This outcome will be evaluated with neuropsychological tests: psychometric hepatic encephalpathy score (PHES) and the critical flicker frequency test (CFF)
No increase in the rate of variceal bleeding and no progression in the number/size of esophageal varices | 3 months
  History taking, hemoglobin measurement, and endoscopy for a detailed description regarding number and size of esophageal varices
Improved ammonia metabolism and decrease in oxidative stress | 3 months
  Ammonia, glutamine, glutamate, and glutamine synthetase determinations, as well as oxidative carbonylation of protein
Improvement in physical capacity and exercise tolerance | 3 months
  Metabolic equivalents (METs) achieved in the treadmill test

CONTACTS AND LOCATIONS:
Overall Officials: Sergio Ponce de Leon-Rosales, M.D., Study Chair — Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran / Universidad Nacional Autonoma de Mexico; Florencia Vargas-Voráckova, MD, Study Chair — Instituto Nacional de Ciencias Médicas y Nutrición Salvador Zubirán/ Universidad Nacional Autónoma de México
Locations (2):
- Mexico (2):
  - Instituto Nacional de Cardiologia Ignacio Chavez, Mexico City, Mexico City
  - Instituto Nacional de Ciencias Medicas y Nutricion Salvador Zubiran, Mexico City, Mexico City

REFERENCES:
- [Derived] Macias-Rodriguez RU, Ilarraza-Lomeli H, Ruiz-Margain A, Ponce-de-Leon-Rosales S, Vargas-Vorackova F, Garcia-Flores O, Torre A, Duarte-Rojo A. Changes in Hepatic Venous Pressure Gradient Induced by Physical Exercise in Cirrhosis: Results of a Pilot Randomized Open Clinical Trial. Clin Transl Gastroenterol. 2016 Jul 14;7(7):e180. doi: 10.1038/ctg.2016.38. PMID 27415618